CLINICAL TRIAL: NCT06122818
Title: Evaluation of Sarcopenia in Patients Receiving Home Health Care
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tuğba Aydın, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstanbulPMRTRHomecare-srcpn
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia; Home Health Care
Keywords: Sarcopenia; home health care
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immobile patients receiving home health care — Demographic characteristics, duration of immobility, sarcopenia presence, thigh circumference , Hand grip strength , bioelectrical impedance analysis

SUMMARY:
The aim in the study is to evaluate the presence of sarcopenia in patients receiving home health care; To evaluate the relationship between sarcopenia and age, disease duration, and cause of immobility. In the literature review, a limited number of studies evaluating sarcopenia in home health patients were found.

DETAILED DESCRIPTION:
Home Health Service is the provision of health services needed by immobile and chronic disease patients in the home environment. The purpose of this service is not to diagnose the patient, but rather to follow up, implement and educate the treatment of the diagnosed patient.

The aim of the study is to evaluate the presence of sarcopenia in patients receiving home health care; To evaluate the relationship between sarcopenia and age, disease duration, and cause of immobility. In the literature review, a limited number of studies evaluating sarcopenia in home health patients were found.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving home health care
2. Being at the mental and physical activity level to be able to perform and complete the tests
3. Being 18-85 years old

Exclusion Criteria:

1) Patients who cannot cooperate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immobile patients receiving home health care
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
handgrip strength | three months
  Handgrip strength will be measured using a hand grip dynamometer. Measurements will be taken 3 times in a sitting position with the elbow flexed to 90° and the wrist in neutral position. The measured maximal grip strength will be recorded as hand grip strength. The measurement will be repeated 3 months after the first measurement
calf circumference | three months
  Calf circumference is an anthropometric measurement that indicates fat free muscle mass and has been considered by the World Health Organization (WHO) the most sensitive index for evaluating the decrease in muscle mass. Calf circumference will be measured with an elastic band over the subject's right leg, both sitting and standing. The measurement will be repeated 3 months after the first measurement
Body Mass Index (BMI) | three months
  BMI will be calculated as weight (kg) divided by height2 (m2). The measurement will be repeated 3 months after the first measurement
Skeletal muscle mass | three months
  Skeletal muscle mass will be evaluated using a multi-frequency body composition analysis device. The measurement will be repeated 3 months after the first measurement

CONTACTS AND LOCATIONS:
Overall Officials: Tugba aydın, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hua N, Zhang Y, Tan X, Liu L, Mo Y, Yao X, Wang X, Wiley J, Wang X. Nutritional Status and Sarcopenia in Nursing Home Residents: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Dec 18;19(24):17013. doi: 10.3390/ijerph192417013. PMID 36554892
- [Background] De Spiegeleer A, Kahya H, Sanchez-Rodriguez D, Piotrowicz K, Surquin M, Marco E, Detremerie C, Hussein D, Hope S, Dallmeier D, Decker G, Hrnciarikova D, Czesak J, Toscano-Rico M, Meza-Valderrama D, Bahat G, Descamps A, Wynendaele E, Elewaut D, Vankova H, Landi F, Benoit F, Gasowski J, Van Den Noortgate N. Acute sarcopenia changes following hospitalization: influence of pre-admission care dependency level. Age Ageing. 2021 Nov 10;50(6):2140-2146. doi: 10.1093/ageing/afab163. PMID 34379741
- [Background] Thompson MQ, Jadczak AD, Yu S, Tucker GR, Visvanathan R. Sarcopenia risk in nursing home residents using SARC-F: FIRST study findings. Geriatr Gerontol Int. 2022 Mar;22(3):206-212. doi: 10.1111/ggi.14327. Epub 2022 Jan 13. PMID 35029041
- [Background] Kamo T, Ishii H, Suzuki K, Nishida Y. Prevalence of sarcopenia and its association with activities of daily living among japanese nursing home residents. Geriatr Nurs. 2018 Sep-Oct;39(5):528-533. doi: 10.1016/j.gerinurse.2018.02.011. Epub 2018 Mar 16. PMID 29555099
- [Background] Fashho E, Ahmed T, Garden G, Readman D, Storey L, Wilkinson L, Wilson G, Slee A. Investigating the prevalence of malnutrition, frailty and physical disability and the association between them amongst older care home residents. Clin Nutr ESPEN. 2020 Dec;40:231-236. doi: 10.1016/j.clnesp.2020.09.014. Epub 2020 Sep 22. PMID 33183542